CLINICAL TRIAL: NCT04307199
Title: Feasibility Study Protocol of a Pragmatic, Randomised Controlled Pilot Trial: Membrane Sweeping to Prevent Post-term Pregnancy: The MILO Study
Brief Title: Membrane Sweeping to Prevent Post-term Pregnancy: The MILO Study
Acronym: MILO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Prof. Declan Devane, Scientific Director, HRB-Trials Methodology Research Network, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NUIreland - MILO
Record Dates: First submitted 2020-01-17; First posted 2020-03-13 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy, Prolonged; Induced; Birth; Pregnancy Related
Keywords: membrane sweep; feasibility study; randomised trial; pilot study; SWAT; pregnancy; induction of labour; post dates; prolonged pregnancy
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Intervention Model Description: Women will initially be randomised in a 2:1 ratio to:
  • Membrane sweep (2) versus no membrane sweep (1).
  Those allocated to the intervention group will then be further randomised in a factorial fashion to A, B, C or D:
  A. Membrane sweep @ 39 weeks' gestation only B. Membrane sweep @ 40 weeks' gestation only C. Membrane sweep @ 39, 40 and 41 weeks' gestation or until onset of labour D. Membrane sweep @ 40 and 41 weeks' gestation or until onset of labour
Who Masked: Outcomes Assessor
Masking Description: Clinicians performing a membrane sweep cannot be blinded and it is not feasible to genuinely blind membrane sweeping for women. Therefore, neither clinicians administering the intervention nor women will be blinded to group assignment. Data will be reviewed by two assessors blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Membrane sweep @ 39 weeks' gestation only
  Interventions: Procedure: Amniotic membrane sweep
- Group B (Experimental): Membrane sweep @ 40 weeks' gestation only
  Interventions: Procedure: Amniotic membrane sweep
- Group C (Experimental): Membrane sweep @ 39, 40 and 41 weeks' gestation or until onset of labour
  Interventions: Procedure: Amniotic membrane sweep
- Group D (Experimental): Membrane sweep @ 40 and 41 weeks' gestation or until onset of labour
  Interventions: Procedure: Amniotic membrane sweep
- Control Group (No Intervention): Women in the control arm will not receive a membrane sweep and will receive usual care (as defined by local hospital protocols and vaginal examination to determine Bishop score only).

INTERVENTIONS:
Procedure: Amniotic membrane sweep — Amniotic membrane sweeping is defined as the manual detachment of the inferior pole of the amniotic membranes from the lower uterine segment. This is performed with consent by a clinician digitally through a circular motion during a vaginal examination. If the cervical os is closed massage of the cervix will be accepted.
  Arms: Group A; Group B; Group C; Group D

SUMMARY:
Multicentre, pragmatic, parallel group, pilot randomised controlled trial with an embedded factorial design.

DETAILED DESCRIPTION:
The primary aim of the MILO study is to inform the optimal design of a future definitive randomised trial to evaluate the effectiveness (including optimal timing and frequency) of membrane sweeping to prevent post-term pregnancy. We will also assess the acceptability and feasibility of the proposed trial interventions to clinicians and women (through focus group interviews).

Methods/Design

Multicentre, pragmatic, parallel group, pilot randomised controlled trial with an embedded factorial design. Pregnant women with a live, singleton fetus ≥ 38 weeks gestation, cephalic presentation, longitudinal lie, intact membranes, English speaking and ≥18 years of age will be randomised in a 2:1 ratio to:

• Membrane sweep versus no membrane sweep

Women allocated randomly to a sweep will then be randomised further (factorial component) to:

* early (from 39 weeks) versus late (from 40 weeks) sweep commencement; and
* a single verses weekly sweep

The proposed feasibility study consists of four work packages i.e., (1) a multicentre, pilot randomised trial, 2) a health economic analysis and 3) a qualitative study (4) a study within the host trial (a SWAT).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women carrying a live singleton fetus ≥ 38 weeks completed gestation.
* (Gestational age will be calculated from the first day of the last menstrual period and an
* ultrasound examination carried out in the 2nd trimester)
* Longitudinal lie
* Cephalic presentation
* Intact amniotic
* ≥ 18 years of age on enrollment

Exclusion Criteria:

* Not able to communicate in english
* contraindications to a vaginal examination
* contraindications to a vaginal birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2020-07-30 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Duration of the recruitment process (approximately 8 months )
  Evaluation of the number and percentage of eligible women who are recruited and randomised to the study. Assessed by study-specific checklists.
Retention | At month 15 approximately
  Evaluation of the number and percentage of eligible women who are randomised, take part in and adhere to the study protocols. Data will be extracted from routinely collected data.
Adherence with the trial interventions. | At month 15 approximately
  Evaluation of adherence with the trial interventions, and reasons for non-compliance assessed by study-specific checklists. Data will be extracted from routinely collected data and focus group interviews with clinicians and participants at six weeks post intervention.
Evaluation of the randomisation process. | At month 15 approximately
  Evaluation of effective allocation of participants to the intervention/control group assessed by study-specific checklists and evaluation of the randomisation protocol throughout the randomisation period.
Evaluation of attrition rates | At month 15 approximately
  Evaluation of attrition rates assessed by study-specific checklists. Data will be extracted from routinely collected data.
Evaluation of the types of attrition | At month 21 approximately
  Evaluation of the types of attrition assessed by case report forms. Data will be extracted from routinely collected data.
Evaluation of the data collection process through study specific checklists | At month 21 approximately
  Evaluated, statistically and narratively, by assessing the completeness of outcome measurements at baseline and postnatal (6 weeks) through study specific checklists. Researchers will manually examine the data collected. They will assess the proportion of complete data collection forms, the quality of data collected and the applicability of this data in facilitating pilot trial outcomes.
Estimate the main effect of individual intervention components and their interactions | At month 21 approximately
  Estimates (with measures of uncertainty) of the main effect of individual intervention components and any interaction effect between the main effects of the embedded factorial design will be assessed and reported using regression analysis.
Evaluation of the data analysis process | At month 21 approximately
  As this is a feasibility study formal hypothesis testing will not be undertaken. Researchers will manually examine the data collected. Evaluation of the data analysis process will be undertaken through the assessment of gaps and limitations to the analysis process measured by study-specific checklist. Findings will be reported through descriptive statistics and graphical summaries.
Evaluation of the EQ5D | At month 21 approximately
  Assessment of the mechanism of, timing of and delivery of the EQ5D through study specific checklists.
Feasibility of cost analyses process through analysis of study specific documentation. | At month 21 approximately
  Assessment of data collection tools to undertake cost effectiveness analysis through study specific documentation. Researchers will manually examine data to assess the mechanism of, timing of and delivery of the cost analysis tools.
Feasibility of the cost effectiveness analyses | At month 21 approximately
  Assessment of the mechanism and utilisation of the incremental cost-effectiveness ratio (ICER), through study specific checklists.

SECONDARY OUTCOMES:
Number of participants achieving a spontaneous onset of labour | From time of randomisation to commencement of spontaneous onset of labour or formal induction of labour or caesarean section (up to 5 weeks)
  Labour which begins spontaneously.
Number of participants who underwent an induction of labour | From time of randomisation to commencement of formal induction of labour (up to 5 weeks).
  Formal induction of labour using pharmacological or surgical methods.
Number of participants achieving a spontaneous vaginal birth | From time of randomisation to birth of baby (up to 5 weeks)
  Spontaneous vaginal birth
Instrumental birth | From time of randomisation to birth of baby (up to 5 weeks)
  Vaginal birth which is assisted with the use of instruments.
Caesarean Section | From time of randomisation to birth of baby (up to 5 weeks)
  Birth which is achieved through the surgical procedure caesarean section.
Post-Partum Haemorrhage ≥ 500mls | From time of birth to 24 hours after the birth of baby.
  Blood loss ≥ 500mls within the first 24 hours of the birth of a baby
Antepartum haemorrhage requiring hospital admission | From 24+0 weeks of pregnancy to birth of baby (up to 18 weeks)
  Bleeding from the genital tract, from 24+0 weeks of pregnancy and before the birth of the baby.
Uterine hyperstimulation with/without fetal heart rate (FHR) changes | From time of randomisation to birth of baby (up to 5 weeks)
  Uterine hyperstimulation defined as uterine tachysystole (more than five contractions per ten minutes for at least twenty minutes) and uterine hypersystole/hypertonicity (a contraction lasting at least two minutes). These may or not be associated with changes in the fetal heart rate pattern (persistent decelerations, tachycardia or decreased short term variability.
Serious maternal death or morbidity | From time of randomisation to six weeks postnatal (up to 11 weeks).
  Serious maternal death or morbidity (e.g. uterine rupture, admission to intensive care unit, septicaemia)
Epidural analgesia | From time of randomisation to birth of baby (up to 5 weeks)
  Introduction of a local anaesthetic into the epidural space of the vertebral canal.
Augmentation of labour | From commencement of established labour to birth of baby (up to 2 days)
  The stimulation of uterine contractions using pharmacologic methods or artificial rupture of membranes to increase their frequency and/or strength following the onset of spontaneous labor or contractions following spontaneous rupture of membranes (ACOG 2014)
Pyrexia in labour | From commencement of established labour to birth of baby (up to 2 days)
  Pyrexia that developed anytime after onset of labour.
Uterine rupture | From time of randomisation to birth of baby (up to 5 weeks)
  All clinically signiﬁcant ruptures of unscarred or scarred uteri. Trivial scar dehiscence noted incidentally at the time of surgery will be excluded
EQ5D-5L | From time of randomisation to six weeks postnatal (up to 11 weeks)
  EuroQol EQ5D-5L survey instrument.
Serious neonatal morbidity | From time of birth of baby to six weeks postnatal.
  e.g. seizures, birth asphyxia defined by trialists, neonatal encephalopathy, disability in childhood, Proven and suspected neonatal sepsis
Apgar score < 7 at five minutes. | From birth of baby to five minutes of life.
  The Apgar score provides an accepted and convenient method for reporting the status of the newborn infant immediately after birth and the response to resuscitation if needed (ACOG 2015).
Cord PH < 7.20 | From birth of infant to collection of cord bloods after delivery of the placenta (an average of 15 minutes)
  Umbilical cord blood gas test.
Neonatal encephalopathy | From time of birth to six weeks postnatal.
  Severity of hypoxic ischaemic encephalopathy assessed using Sarnat staging; i)Stage 1 (mild): hyper-alertness, hyper-reflexia, dilated pupils, tachycardia, absence of seizures; ii)Stage 2 (moderate): lethargy, hyper-reflexia, miosis, bradycardia, seizures, hypotonia with weak suck and Moro reflexes; iii)Stage 3 (severe): stupor, flaccidity, small to mid-position pupils which react poorly to light, decreased stretch reflexes, hypothermia and absent Moro reflex.
Perinatal death | From time of randomisation to seven completed days after birth of baby (up to 6 weeks)
  The perinatal period is defined as "commences at 22 completed weeks (154 days) of gestation and ends seven completed days after birth of baby."
Admission to neonatal intensive care unit or equivalent | From time of birth to six weeks postnatal.
  Admission of infant to neonatal intensive care unit or equivalent
Length of time from membrane sweep to birth of baby. | From time of membrane sweep to birth of baby (up to 4 weeks)
  Length of time from membrane sweep to birth of baby .
Length of time from formal induction of labour to birth of baby. | From time of formal induction of labour to birth of baby (up to 2 weeks)
  Length of time from formal induction of labour to birth of baby.
Overall length of maternal hospital stay | From time of randomisation to six weeks postnatal (up to 11 weeks).
  Overall length of maternal hospital stay
Length of infant stay in neonatal intensive care unit or equivalent | From time of birth to six weeks postnatal.
  Length of infant stay in neonatal intensive care unit or equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Declan Devane, PhD, Principal Investigator — National University of Ireland, Galway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finucane EM, Biesty L, Murphy D, Cotter A, Molloy E, O'Donnell M, Treweek S, Gillespie P, Campbell M, Morrison JJ, Alvarez-Iglesias A, Gyte G, Devane D. Feasibility study protocol of a pragmatic, randomised controlled pilot trial: membrane sweeping to prevent post-term pregnancy-the MILO Study. Trials. 2021 Feb 2;22(1):113. doi: 10.1186/s13063-021-05043-9. PMID 33531062